CLINICAL TRIAL: NCT04646655
Title: Enoxaparin at Prophylactic or Therapeutic Doses With Monitoring of Outcomes in Subjects Infected With COVID-19: a Pilot Study on 300 Cases Enrolled at ASST-FBF-Sacco
Brief Title: Enoxaparin at Prophylactic or Therapeutic Doses in COVID-19
Acronym: EMOS-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Massimo Arquati (Unknown); Riccardo Colombo (Unknown); Umberto Russo (Unknown); Manuela Nebuloni (Unknown); Spinello Antinori (Unknown)
Responsible Party: Principal Investigator, Maddalena Alessandra Wu, Principal Investigator, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLS-02COVID19/2020
Record Dates: First submitted 2020-11-22; First posted 2020-11-30 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Covid19; Thrombosis
Keywords: COVID.19; Thrombosis; Enoxaparin; Outcome; Respiratory failure; D-dimer; Venous compression ultrasound
MeSH Terms: conditions — COVID-19; Thrombosis; Respiratory Insufficiency | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxaparin at prophylactic dose (Active Comparator): Enoxaparin at prophylactic dose: standard 4.000 IU QD via subcutaneous injection (6000 IU if body weight>100 kg)
  Interventions: Drug: Enoxaparin
- Enoxaparin at therapeutic dose (Experimental): Enoxaparin at therapeutic dose : 70 U/Kg b.i.d. (every 12 h)
  In order to easily calculate the correct therapeutic dose of enoxaparin for each patient, a simplified categorization will be applied, as follows:
  * weight < 65 Kg: 4.000 IU b.i.d. (every 12 h)
  * weight ≥ 65 Kg: 6.000 IU b.i.d. (every 12 h)
  * weight ≥ 100 Kg: 8.000 IU b.i.d. (every 12 h) The most appropriate dose will be evaluated in patients with creatinine clearance between 30 and 50 ml/min
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — subcutaneous injections
  Other Names: Clexane

SUMMARY:
SINGLE CENTER PHASE III INTERVENTIONAL RANDOMIZED CONTROLLED TRIAL comparing efficacy and safety of enoxaparin at prophylactic dose (standard treatment) and enoxaparin at therapeutic dose (OFF-LABEL treatment) in 300 COVID-19 infected patients with moderate-severe respiratory failure (PaO2/FiO2<250) and/or increased D-dimer levels enrolled in different Units (Infectious disease, Internal Medicine, Emergency Medicine, Pneumology) of Azienda Socio Sanitaria Territoriale Fatebenefratelli Sacco (ASST-FBF-SACCO).

DETAILED DESCRIPTION:
Patients with COVID-19 are at high risk of developing a venous thromboembolism (VTE) and it is essential that effective thromboprophylaxis with parenteral drugs (LMWH, UFH) is considered for all patients admitted to hospital especially in case of severe pneumonia.

The aim of the study is the evaluation of efficacy and safety of enoxaparin at prophylactic dose (standard treatment) as compared to enoxaparin at therapeutic dose (OFF-LABEL treatment) in 300 COVID-19 infected patients with moderate-severe respiratory failure (PaO2/FiO2<250) and/or increased D-dimer levels.

After the admission to different Units (Infectious disease, Internal Medicine, Emergency Medicine, Pneumology), enoxaparin at prophylactic dose (standard of care) will be prescribed to all patients.

The randomization of the single patient will be made when the the inclusion criteria (PaO2/FiO2 <250 and/or D-dimer >2000 ng/) will be satisfied. Patients with increased bleeding risk will be excluded (exclusion criteria).

Patients will be divided into two arms:

* arm A: enoxaparin at prophylactic dose (standard 4.000 IU; 6000 UI if body weight>100 kg)
* arm B: enoxaparin at therapeutic dose (70 U/Kg b.i.d. every 12 h)

In both arms, enoxaparin treatment will be monitored clinically and with first and second line laboratory tests Venous compression ultrasound (CUS) will be performed at admission and after 7 days in case of a first negative exam and elevated D-Dimer levels, to rule out deep vein thrombosis.

Enoxaparin at prophylactic dose (4000 IU) will be maintained in all patients for 4 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 related pneumonia with moderate-severe respiratory failure (PaO2/FiO2<250) and/or markedly increased D-dimer level (>2000 ng/mL)
* Signed informed consent

Exclusion Criteria:

* age < 18 and > 80 yrs
* history of bleeding (peptic ulcer, esophageal varices, cerebral aneurysm, cancer at high risk of bleeding, cirrhosis, hemorrhagic stroke < 1 year)
* thrombocytopenia (<100 x109/L)
* anemia (Hb < 8 g/dl)
* coagulation abnormalities (PT e/o aPTT > 1.5; fibrinogen < 150 mg/dl)
* consumption coagulopathy (ISTH criteria) [15, 16]
* deep vein thrombosis or pulmonary embolism
* dual antiplatelet therapy
* ongoing anticoagulant therapy
* allergic reaction to LMWH
* previous heparin-induced thrombocytopenia
* major surgery < 1 month; neurosurgery <3 months; eye surgery <3 months
* pregnancy
* arterial hypertension (SBPS>160 mm Hg; DBP>100 mm Hg)
* renal failure (creatinine clearance 30 ml/min)
* ICU admission or endotracheal intubation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 30 days from enrollment
  Mortality registered during the time frame
Progression of respiratory failure | 30 days from enrollment
  Progression of respiratory failure defined as duration of continuous positive pressure ventilation (CPAP)
Progression of respiratory failure | 30 days from enrollment
  Progression of respiratory failure defined as percentage of patients admitted to ICU
Progression of respiratory failure | 30 days from enrollment
  Progression of respiratory failure defined as percentage of patients undergoing oro-tracheal intubation
Number of major bleeding episodes | up to 6 months from randomization
  Major bleeding (ISTH criteria) and/or clinically relevant non-major bleeding

SECONDARY OUTCOMES:
Respiratory function improvement | at 72 hours
  Amelioration of the respiratory function defined as a PaO2/FiO2 increase > 300 and / or respiratory rate (RR) < 20 breaths per min
Respiratory function improvement | 1 week from randomization
  Amelioration of the respiratory function defined as a PaO2/FiO2 increase > 300 and / or respiratory rate (RR) < 20 breaths per min
Number of major cardiovascular events | 6 months from randomization
  numbers of myocardial infarction and stroke within the time frame
Deep Vein Thrombosis | 6 months from randomization
  Numbers of Deep Vein Thrombosis at CUS examination within the time frame

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena A Wu, M.D., Principal Investigator — ASST Fatebenefratelli Sacco
Locations (1):
- ASST Fatebenefratelli Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han H, Yang L, Liu R, Liu F, Wu KL, Li J, Liu XH, Zhu CL. Prominent changes in blood coagulation of patients with SARS-CoV-2 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1116-1120. doi: 10.1515/cclm-2020-0188. PMID 32172226
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] McGonagle D, Sharif K, O'Regan A, Bridgewood C. The Role of Cytokines including Interleukin-6 in COVID-19 induced Pneumonia and Macrophage Activation Syndrome-Like Disease. Autoimmun Rev. 2020 Jun;19(6):102537. doi: 10.1016/j.autrev.2020.102537. Epub 2020 Apr 3. PMID 32251717
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Background] Iba T, Nisio MD, Levy JH, Kitamura N, Thachil J. New criteria for sepsis-induced coagulopathy (SIC) following the revised sepsis definition: a retrospective analysis of a nationwide survey. BMJ Open. 2017 Sep 27;7(9):e017046. doi: 10.1136/bmjopen-2017-017046. PMID 28963294
- [Background] Young E. The anti-inflammatory effects of heparin and related compounds. Thromb Res. 2008;122(6):743-52. doi: 10.1016/j.thromres.2006.10.026. Epub 2007 Aug 28. PMID 17727922
- [Background] Poterucha TJ, Libby P, Goldhaber SZ. More than an anticoagulant: Do heparins have direct anti-inflammatory effects? Thromb Haemost. 2017 Feb 28;117(3):437-444. doi: 10.1160/TH16-08-0620. Epub 2016 Dec 15. PMID 27975101
- [Background] Mousavi S, Moradi M, Khorshidahmad T, Motamedi M. Anti-Inflammatory Effects of Heparin and Its Derivatives: A Systematic Review. Adv Pharmacol Sci. 2015;2015:507151. doi: 10.1155/2015/507151. Epub 2015 May 12. PMID 26064103
- [Background] Thachil J. The versatile heparin in COVID-19. J Thromb Haemost. 2020 May;18(5):1020-1022. doi: 10.1111/jth.14821. Epub 2020 Apr 27. No abstract available. PMID 32239799
- [Background] Milewska A, Zarebski M, Nowak P, Stozek K, Potempa J, Pyrc K. Human coronavirus NL63 utilizes heparan sulfate proteoglycans for attachment to target cells. J Virol. 2014 Nov;88(22):13221-30. doi: 10.1128/JVI.02078-14. Epub 2014 Sep 3. PMID 25187545
- [Background] Barrett CD, Moore HB, Yaffe MB, Moore EE. ISTH interim guidance on recognition and management of coagulopathy in COVID-19: A comment. J Thromb Haemost. 2020 Aug;18(8):2060-2063. doi: 10.1111/jth.14860. Epub 2020 Jun 14. No abstract available. PMID 32302462
- [Background] Wada H, Thachil J, Di Nisio M, Mathew P, Kurosawa S, Gando S, Kim HK, Nielsen JD, Dempfle CE, Levi M, Toh CH; The Scientific Standardization Committee on DIC of the International Society on Thrombosis Haemostasis. Guidance for diagnosis and treatment of DIC from harmonization of the recommendations from three guidelines. J Thromb Haemost. 2013 Feb 4. doi: 10.1111/jth.12155. Online ahead of print. PMID 23379279
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170